CLINICAL TRIAL: NCT01107041
Title: Technology Assisted Intervention for the Treatment and Prevention of Depression
Brief Title: Mobile Phone Sensing and Outreach as Adjuncts to Internet-Based Behavioral Intervention for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, David Mohr, Director, Center for Behavioral Intervention Technologies; Professor, Department of Preventive Medicine, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P20MH090318 STU00021825; P20MH090318 (NIH)
Record Dates: First submitted 2010-04-19; First posted 2010-04-20 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2015-10

CONDITIONS: Depression
Keywords: Depression; Technology Assisted; Mobile Phone
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: This study is collecting phone sensor data and ecological momentary assessment data to try to develop algorithms that can passively detect behavioral patterns in participants
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mobilyze! (Experimental)
  Interventions: Behavioral: Mobilyze!

INTERVENTIONS:
Behavioral: Mobilyze! — Mobilyze! delivers behavioral intervention for depression via a mobile phone, interactive website, and e-mail.

SUMMARY:
Investigators are evaluating the use of phone sensor data to estimate behavior, depression and anxiety.

DETAILED DESCRIPTION:
Investigators are evaluating the use of phone sensor data to estimate behavior, depression and anxiety. Participants will include people who are high on depression, high on anxiety, hight on both depression and anxiety, and health controls. Particpants will load software on their phones that collects phone sensor data, and obtains self report on sleep, mood, and social contacts. Data will be collected for at least 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* PHQ-9 score 10 or higher
* Has an e-mail account, computer, and broadband access to the Internet
* Familiarity with mobile phones and is within a cellular network range the majority of the day.
* Is able to speak and read English.
* Is at least 19 years of age.

Exclusion Criteria:

* Hearing or voice impairment preventing participation in psychotherapy.
* Visual impairment that would prevent use of the website, mobile phone application, and assessment materials.
* Has any psychiatric condition for which participation in a clinical trial of psychotherapy may be either inappropriate or dangerous (e.g., psychotic disorders, bipolar disorders, dissociative disorders, etc.).
* Planning to be out of town or unavailable for intervention for 1 or more weeks during the scheduled study participation.
* Exhibits severe suicidality, including ideation, plan, and intent.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2010 (Actual)
Dates: Start 2014-12; Primary Completion 2016-02 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Depression, as assessed the Patient Health Questionnaire-9 | Baseline, Weeks 2-6

SECONDARY OUTCOMES:
Positive Affect (PANAS - Positive Affect Scale) | Baseline, Weeks 2-6
Anxiety (GAD-7) | Baseline, Weeks 2-6

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Burns MN, Begale M, Duffecy J, Gergle D, Karr CJ, Giangrande E, Mohr DC. Harnessing context sensing to develop a mobile intervention for depression. J Med Internet Res. 2011 Aug 12;13(3):e55. doi: 10.2196/jmir.1838. PMID 21840837
- See also: MedlinePlus — http://www.nlm.nih.gov/medlineplus/
- See also: Depression at MedlinePlus Site — http://www.nlm.nih.gov/medlineplus/depression.html
- See also: Mental Health at MedlinePlus Site — http://www.nlm.nih.gov/medlineplus/mentalhealth.html